CLINICAL TRIAL: NCT03835247
Title: Physician-Nurse and Nurse-Nurse Collaboration in Different Hospitals: An Example From Turkey
Brief Title: Physician-Nurse and Nurse-Nurse Collaboration
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Ebru ŞAHİN, Asisstant professor, Ordu University
Other Study IDs: collaboration
Record Dates: First submitted 2019-02-07; First posted 2019-02-08 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Nurse
Keywords: physician-nurse collaboration; nurse-nurse collaboration

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was carried out to determine the level of collaboration and the factors affecting its between physicians-nurses and nurses-nurses working in different hospitals.

DETAILED DESCRIPTION:
Collaboration is a broad concept with different definitions in the literature. Researches on physician-nurse collaboration and nurse-nurse collaboration has shown that improves the quality of patient care; reduces the medical errors; affects the job satisfaction positively and decreases the intention to quit in the international literature. In the light of this information, the study was planned to determine the level of collaboration and the factors affecting its between physicians-nurses and nurses-nurses working in different hospitals. Research is a cross-sectional study. The study is planned the 500 nurses working in six hospitals in Ordu/Turkey on January 3-12 February 2019. Descriptive questionnaire form, Jefferson Scale of Physician-Nurse Collaboration (JSAPNC) and nurse-nurse collaboration scale will be used in the study.

ELIGIBILITY:
Inclusion Criteria:

* nurse
* working experiences at least 6 months
* working full time.

Exclusion Criteria

* working experiences less than 6 months
* head-nurses

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 500 nurses working in six hospitals.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-02-12 (Estimated); Study Completion 2019-02-19 (Estimated)

PRIMARY OUTCOMES:
Descriptive questionnaire form, | 2 minutes
  Descriptive questionnaire form includes nurse's age, gender, education, clinical experiences and hospital types etc.
Jefferson Scale of Physician-Nurse Collaboration | 3 minutes
  The scale includes 15 question about physician and nurse collaboration.
nurse-nurse collaboration scale | 5 minutes
  The scale includes 35 question about nurse and nurse collaboration.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Sahin, Phd, Principal Investigator — Ordu University
Locations (1):
- Hospitals, Ordu, Altınordu, Turkey (Türkiye)

REFERENCES:
- [Derived] Sahin E, Catiker A, Ozdil K. Physician-Nurse and Nurse-Nurse Collaboration From the Perspective of Nurses: A Cross-Sectional Study. J Nurses Prof Dev. 2023 Jan-Feb 01;39(1):E8-E17. doi: 10.1097/NND.0000000000000779. Epub 2021 Sep 7. PMID 34516465